CLINICAL TRIAL: NCT04547569
Title: Somesthesic Role of the Ventro-lateral Prefrontal Cortex in Speech Motor Learning fMRI Study
Brief Title: Somesthesic Role of the Ventro-lateral Prefrontal Cortex in Speech Motor Learning
Acronym: BRAVA²
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other); GIPSA-LAB (Other); McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC18.173
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Speech; Motor Activity
MeSH Terms: conditions — Speech; Motor Activity | interventions — Speech, Alaryngeal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adaptation to altered auditory feedback (Experimental): fMRI measurement of brain activity during speech production under altered auditory feedback
  Interventions: Behavioral: Speech adaptation; Other: fMRI
- Speech production (Experimental): fMRI measurement of brain activity during normal speech production
  Interventions: Other: fMRI; Behavioral: Speech production
- Vibrotactile discrimination (Experimental): fMRI measurement of brain activity during a vibrotactile discrimination task
  Interventions: Behavioral: Vibrotactile Discrimination; Other: fMRI

INTERVENTIONS:
Behavioral: Speech adaptation — Sensorimotor adaptation in speech
  Arms: Adaptation to altered auditory feedback
Behavioral: Vibrotactile Discrimination — Vibrotactile Discrimination
  Arms: Vibrotactile discrimination
Other: fMRI — fMRI measurement of brain activity
Behavioral: Speech production — Speech production task
  Arms: Speech production

SUMMARY:
These studies test the hypothesis that frontal areas of the brain participate in the cortical networks involved in the somotosensory processing that happens during speech motor learning.

DETAILED DESCRIPTION:
This work aims to study the role of sensory systems in human motor learning and specifically addresses the involvement of somatosensory cortical networks in motor learning of speech. Previous studies in the literature have highlighted the plasticity of cortical sensory networks, notably the primary and secondary somatosensory cortex and the ventral premotor cortex, during motor learning tasks. The present project focuses on the somatosensory region with connections to the sensorimotor regions of the frontal and parietal cortex. We propose to use neuroimaging (fMRI), in order to verify which areas in the prefrontal cortex are part of the sensorimotor network used in the learning of speech motor tasks in humans. Subjects will be tested in the fMRI scanner while performing either a behavioral task in which the auditory feedback of their own speech is altered or while performing a vibrotactile discrimination task.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed subjects
* Subjects fluent in French
* Signed informed consent
* Affiliation to or beneficiary of a Social Security scheme

Exclusion Criteria:

* Left-handed subjects
* Criteria for contraindications to protocol fMRI scans
* Existence of a severe general condition: cardiac, respiratory, hematological, renal, hepatic, cancerous.
* Hearing, language (including dyslexia), neurological or psychiatric disorders.
* Participation in other ongoing intervention research protocols with exclusionary period or within the previous week
* Drug treatment likely to modulate brain activity: benzodiazepines, antidepressants, neuroleptics, lithium, etc.
* Protected persons referred to in articles L1121 5 to L1121 8 of the French CSP:

  * Pregnant women, parturients, nursing mothers,
  * Persons deprived of liberty by a judicial or administrative decision,
  * Persons under psychiatric care,
  * Individuals admitted to a health or social institution for purposes other than research,
  * Minors,
  * Persons over the age of majority who are subject to a legal protection measure or who are unable to express their consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Motor Learning | Performance as measured at the end of learning (during the 1h30 scanner session)
  Learning is assessed as percentage change in speech sounds (speech formant frequencies) relative to baseline.
Brain activity | 1h30 scanner session
  Brain activity are measure by the BOLD signal during both task-based and resting-state blocks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France